CLINICAL TRIAL: NCT02448732
Title: Exploratory Clinical Trials of ACM-1 in the Treatment of Ophthalmological Neovascular Diseases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qianying Gao, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sun Yat-sen Un
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Neovascularization, Pathologic
Keywords: ACM-1; intravitreal injection; neovascularization
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACM-1 team (Experimental): intravitreal injection with 50ul ACM-1 at a concentration of 1600ug/ml
  Interventions: Drug: ACM-1

INTERVENTIONS:
Drug: ACM-1 — intravitreal injection with 50ul ACM-1 at a concentration of 1600ug/ml

SUMMARY:
The purpose of this study is to investigate the role of intravitreal injection of anti-vascular endothelial growth factor (VEGF) therapy in prevention and control of ophthalmological neovascular diseases, in order to find a new strategy of treatment for ophthalmological neovascular diseases

DETAILED DESCRIPTION:
Ophthalmological neovascular disease is one of the major causes of blindness in ocular diseases. Up to now, the major treatment strategies include: anti-VEGF therapy, laser therapy and surgery. Clinical treatment have revealed that intravitreal injection of anti-VEGF can effectively restrain neovascularization. Nevertheless, it requires repeated injections, may result in various complications, and may be ineffective in some patients. Therefore, it is necessary to find out other targets which causes retinal neovascularization, in order to find more effective treatments for patients who fail to respond to anti-VEGF therapy. Previous researches have shown that herb monomer (ACM-1) was effective in inhibiting leakage of retinal vessels and neovascularization. So in this study, patients with ophthalmological neovascular diseases will be treated with intravitreal injection of ACM-1, in order to investigate the role of intravitreal injection of ACM-1 therapy in prevention and control of ophthalmological neovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

1. age range from 18 to 75 years old
2. without light perception (NLP)
3. A large number of iris or retinal neovascularizations, neovascular glaucoma who needs cyclophotocoagulation or enucleation of eyeball
4. The best corrected visual acuity of the contralateral eye is better than 0.05
5. Follow-up for more than six months
6. Volunteer for this project and sign the informed consent

Exclusion Criteria:

1. The best corrected visual acuity of the contralateral eye is lower than 0.05
2. Severe systemic disease or other surgical contraindication
3. history of antiangiogenic therapy within one month
4. Ocular neovascularization was caused by other reasons,such as endophthalmitis
5. history of joining in drug clinical trial within one month(except for vitamins and minerals)
6. pre-menopausal women who do not use birth control
7. people are currently being treated for systemic infections
8. Allergic to fluorescein
9. hypertension(SBP is higher than 140mmHg)
10. hepatic renal dysfunction
11. History of drug abuse or alcoholism
12. other situation which will impede the clinical trial, as such depressive disorder
13. the compliance is too poor to finish the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
fluorescence fundus angiography | 6 months after treatment

SECONDARY OUTCOMES:
intra-ocular pressure | 6 months after treatment
optical coherence tomography | 6 months after treatment
  change in central retinal/lesion thickness (CR/LT) and the mean decrease in thickness at the foveal center > 100 um or >20% center
Retinal Oximetry | 6 months after treatment
blood pressure | at admission, 1 day ,3days,1 week, 1month ,3moths and 6 months after treatment
ocular inflammatory response | at admission, 1 day ,3days,1 week, 1month ,3moths and 6 months after treatment
morphological changes of the anterior segment | at admission, 1 day ,3days,1 week, 1month ,3moths and 6 months after treatment
Corneal Endothelium Cell Counter | at admission, 1 day ,3days,1 week, 1month ,3moths and 6 months after treatment
adverse event | at admission, 1 day ,3days,1 week, 1month ,3moths and 6 months after treatment
morphological changes of the posterior segment | at admission, 1 day ,3days,1 week, 1month ,3moths and 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qianying Gao, PHD, Principal Investigator — State Key Laboratory of Ophthalmology,Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- State Key Laboratory of Ophthalmology,Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Adatia FA, Luong M, Munro M, Tufail A. The other CNVM: a review of myopic choroidal neovascularization treatment in the age of anti-vascular endothelial growth factor agents. Surv Ophthalmol. 2015 May-Jun;60(3):204-15. doi: 10.1016/j.survophthal.2014.10.002. Epub 2014 Nov 5. PMID 25890624